CLINICAL TRIAL: NCT02552732
Title: Nasal High Flow (NHF) Therapy Use Following Hospitalization for an Exacerbation of COPD: A Feasibility Study
Brief Title: Nasal High Flow Therapy 30 Day Readmission Study
Acronym: N3ADS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to change in business of US site.
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Medical Research Institute of New Zealand (Other); Alana Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIA138
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NHF with or without Oxygen (Experimental): NHF with or without oxygen will be delivered to COPD patients using myAIRVO™ 2 for 30 days post hospital discharge
  Interventions: Device: NHF with or without Oxygen

INTERVENTIONS:
Device: NHF with or without Oxygen — NHF using myAIRVO™ 2 will be set at 25L/min at 37°C. However, all participants are able to lower the delivered temperature to 34°C.

SUMMARY:
The aim of this feasibility study is to provide data for a subsequent randomized controlled trial to investigate if patient outcomes will be improved after an acute COPD exacerbation using domiciliary nasal high flow therapy (NHF) compared to standard care. This feasibility study will investigate the following: process, resources, management and scientific aspects of delivering NHF as an adjunct therapy in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male and female
* Admitted to the respiratory ward(s) of either recruiting hospitals with AECOPD as the primary diagnostic reason for admission.

Exclusion Criteria:

* Given a new home oxygen therapy prescription during the current hospital admission
* The investigator believes the participant or their care giver will be unable to safely use the myAIRVO 2 device following discharge
* They have any other condition which, at the investigator's discretion, is believed may present a safety risk or impact the feasibility of the study or the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fingleton, MBChB, Principal Investigator — Medical Research Institute of New Zealand
Locations (2):
- Alana HealthCare, Liverpool, New York, United States
- Medical Research Institute of New Zealand, Wellington, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- NHF With or Without Oxygen: Patients with or without an existing Oxygen prescription will receive NHF using myAIRVO™ 2.
  NHF with supplemental Oxygen will be given to participants with an oxygen prescription using myAIRVO™ 2: NHF will be set at 25L/min at 37°C. However, all participants are able to lower the delivered temperature to 34°C.
  NHF without supplemental Oxygen will be given to participants who do not have an oxygen prescription using myAIRVO™ 2: NHF will be set at 25L/min at 37°C. However, all participants are able to lower the delivered temperature to 34°C.
Period: Overall Study
Arm/Group | NHF With or Without Oxygen
Started | 29
Used Device | 23
Completed Week 1 | 21
Completed Week 2 | 20
Completed Week 3 | 19
Completed Week 4 | 19
Completed Day 1 and Day 31 Spirometry | 12
Completed | 19
Not Completed | 10
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Day 1 SpO2 > 96% | 1
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.34 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  NZ European | 16
  Maori | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  New Zealand | 20

OUTCOME MEASURES:

1. Primary Outcome: NHF Use for 30 Days Following Discharge After AECOPD
Description: Use will be expressed as hours of myAIRVO 2 use per day over 30 days, as obtained by myAIRVO 2 electronic monitoring
Time Frame: 30 days after hospital discharge
Population: NHF use for 30 days following discharge after AECOPD. Use will be expressed as hours of myAIRVO 2 use per day over 30 days, as obtained by myAIRVO 2 electronic monitoring.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
hours per day | 2.6560 (2.4137)

2. Secondary Outcome: Percentage of Days of Use, Adjusted for Number of Days With myAIRVO 2 at Home
Time Frame: 30 days after hospital discharge
Measure: Number; unit: percentage of days of use
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
percentage of days of use | 57.6

3. Secondary Outcome: Average Use Per Day of the myAIRVO 2 During Week 1
Time Frame: First week after hospital discharge
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 21
hours per day | 3.0319 (3.7065)

4. Secondary Outcome: Average Use Per Day of the myAIRVO 2 During Week 2
Time Frame: Second week after hospital discharge
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 20
hours per day | 1.7715 (2.236)

5. Secondary Outcome: Average Use Per Day of the myAIRVO 2 During Week 3
Time Frame: Third week after hospital discharge
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 19
hours per day | 2.0447 (2.4633)

6. Secondary Outcome: Average Use Per Day of the myAIRVO 2 During Week 4
Time Frame: Fourth week after hospital discharge
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 19
hours per day | 2.22 (2.69)

7. Secondary Outcome: Average Use Per Day on Days of myAIRVO 2 Use
Time Frame: 30 days after hospital discharge
Measure: Mean (Standard Deviation); unit: hours per day on days of myAIRVO 2 use
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
hours per day on days of myAIRVO 2 use | 3.4326 (3.4917)

8. Secondary Outcome: Number of Participants Using Home Oxygen
Time Frame: At study entry
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
Participants | 7

9. Secondary Outcome: Number of Participants Who Reported Having Changed the myAIRVO 2 Flow Settings From the Initial Flow and the Corresponding Reduction in Flow
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
Participants | 5

10. Secondary Outcome: Number of Participants Who Where Screened But Were Excluded From Enrollment
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
Participants | 0

11. Secondary Outcome: Number of Participants Who Reported Having Changed the myAIRVO 2 Temperature Setting From the Initial Setting
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
Participants | 9

12. Secondary Outcome: Number of Participants Who Withdrew From Study After Enrollment, up to 30 Days
Description: Number of participants who withdrew from study after enrollment, up to 30 days
Time Frame: At study completion
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
Participants | 10

13. Secondary Outcome: Number of Participants With at Least One Hospital Readmission Within 30 Days of Discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
Participants | 2

14. Secondary Outcome: Reasons for Hospital Admissions
Description: AECOPD, other respiratory cause or other cause
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 2
Participants
  AECOPD | 2
  Other Respiratory | 0
  Non-respiratory | 0

15. Secondary Outcome: In Those That Had at Least One Hospital Readmission: Number of Readmissions
Time Frame: 30 days after hospital discharge
Measure: Number; unit: readmission/participant
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 2
readmission/participant | 1

16. Secondary Outcome: In Those That Had at Least One Hospital Readmission: Time to First Hospital Readmission
Time Frame: 30 days after hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 2
days | 26 (0)

17. Secondary Outcome: In Those That Had at Least One Hospital Readmission: Hospital Readmission Length
Time Frame: 30 days after hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 2
days | 1 (0)

18. Secondary Outcome: Number of Participants With at Least One ED Visit Within 30 Days of Discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 23
Participants | 1

19. Secondary Outcome: Reason for ED Visits
Description: ED visit due to AECOPD
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 1
Participants | 1

20. Secondary Outcome: Number of Participants With at Least One GP Visit Within 30 Days of Discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
Participants | 4

21. Secondary Outcome: LACE Index for Hospital Admissions
Description: The LACE Index is a scoring tool for assessing the likelihood of readmission or death within 30 days of discharge. It is based of 4 parameters: length of stay (L), acuity of the admission (A), co-morbidities (C), number of Emergency Department visits within the last 6 months (E). Sub scores for each parameter are summed to give a LACE score ranging from 1 to 19. A score of 0 to 4 = Low; 5 to 9 = Moderate; and a score of ≥ 10 = High risk of readmission.
Time Frame: 30 days after hospital discharge
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 29
scores on a scale | 11.069 (1.4188)

22. Secondary Outcome: FEV1 at Day 1 and 31
Description: FEV1 change from day 1 to day 31
Time Frame: 1st and 31st day after hospital discharge
Measure: Mean (Standard Deviation); unit: litres per min
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 12
litres per min | 0.0042 (0.1973)

23. Secondary Outcome: SVC(in) at Day 1 and 31
Description: Slow Vital Capacity (inspiratory) change from day 1 to day 31
Time Frame: 1st and 31st day after hospital discharge
Measure: Mean (Standard Deviation); unit: litres per min
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 12
litres per min | 0.0027 (0.393)

24. Secondary Outcome: FVC Change From Day 1 to Day 31
Time Frame: 1st and 31st day after hospital discharge
Measure: Mean (Standard Deviation); unit: litres per min
Arm/Group | NHF With or Without Oxygen
Number analyzed (Participants) | 12
litres per min | 0.075 (0.3306)

ADVERSE EVENTS:
Time Frame: Over 31 days (1 month)
Arm/Group | NHF With or Without Oxygen
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NHF With or Without Oxygen (N=29)
General unwellness/tired (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oral thrush (Infections and infestations) | 1 (1)
AECOPD (Respiratory, thoracic and mediastinal disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT02552732/Prot_SAP_000.pdf